CLINICAL TRIAL: NCT01281254
Title: A Phase 3, Randomized, Double-Blind Trial of Pegylated Liposomal Doxorubicin (PLD) Plus AMG 386 or Placebo in Women With Recurrent Partially Platinum Sensitive or Resistant Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: AMG 386 (Trebananib) in Ovarian Cancer (TRINOVA-2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closure of long term follow up (LTFU) and study earlier than previously outlined in the protocol as no beneficial information gained from continuing LTFU.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20060517; 2009-017946-30 (EudraCT Number); ENGOT-ov-6; TRINOVA-2 (Other: Amgen, Inc); 20060517 (Other: Amgen. Inc.)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cancer
Keywords: Fallopian tube cancer; Primary peritoneal cancer; AMG386; Pegylated Liposomal Doxorubicin; Recurrent epithelial ovarian cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — trebananib; 1-dodecylpyridoxal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo plus PLD (Placebo Comparator): Arm B: PLD 50 mg/m2 IV every 4 weeks (Q4W) and blinded AMG 386 placebo IV weekly (QW)
  Interventions: Drug: Placebo plus PLD
- AMG386 plus PLD (Experimental): Arm A: PLD 50 mg/m2 IV every 4 weeks (Q4W) and blinded AMG 386 15 mg/kg IV weekly (QW)
  Interventions: Drug: AMG386 plus PLD

INTERVENTIONS:
Drug: AMG386 plus PLD — AMG 386 is a first in class investigational anti angiogenic drug that provides potent and selective inhibition of angiopoietins. AMG 386 is designed to inhibit angiogenesis by sequestering Ang1 and Ang2, thereby preventing their interaction with the Tie2 receptor. Pegylated Liposomal Doxorubicin (Doxil/Caelyx) is a preparation of doxorubicin in a liposome that contains surface-grafted segments of the hydrophilic polymer methoxypolyethylene glycol associated with prolonged pharmacokinetics of the free drug. PLD 50 mg/m2 IV every 4 weeks (Q4W) and blinded AMG 386 15 mg/kg IV weekly (QW)
  Arms: AMG386 plus PLD
Drug: Placebo plus PLD — Pegylated Liposomal Doxorubicin (Doxil/Caelyx) is a preparation of doxorubicin in a liposome that contains surface-grafted segments of the hydrophilic polymer methoxypolyethylene glycol associated with prolonged pharmacokinetics of the free drug.
  PLD 50 mg/m2 IV every 4 weeks (Q4W) and blinded AMG 386 placebo IV weekly (QW)
  Arms: Placebo plus PLD

SUMMARY:
To determine if AMG 386 plus pegylated liposomal doxorubicin (PLD) is superior to placebo plus PLD as measured by progression-free survival (PFS)

The hypothesis for this study is that AMG 386 plus PLD will prolong PFS compared to placebo plus PLD in women with recurrent partially platinum sensitive or resistant epithelial ovarian, primary peritoneal or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented invasive epithelial ovarian, primary peritoneal, or fallopian tube cancer
* Radiographically documented disease progression either on or following the last dose of the prior regimen for epithelial ovarian, primary peritoneal, or fallopian tube cancer
* Subjects must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound.
* Female 18 years of age or older at the time the written informed consent is obtained
* Adequate organ and hematological function

Exclusion Criteria:

* Subjects who have received more than 3 previous regimens of anti cancer therapy for epithelial ovarian, primary peritoneal or fallopian tube cancer
* Subjects treated with prior pegylated liposomal doxorubicin (PLD) or any anthracycline-based or mitoxantrone-based chemotherapy
* Subjects with primary platinum-refractory disease
* Subjects with platinum-free interval (PFI) > 12 months from their last platinum based therapy
* History of central nervous system metastasis
* Major surgery within 28 days prior to randomization or still recovering from prior surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-04-18 (Actual); Primary Completion 2014-08-29 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
To determine if AMG 386 plus PLD is superior to placebo plus PLD as measured by progression-free survival, defined as the time from randomization to the earliest of the dates of first radiologic disease progression per RECIST 1.1 with modifications | Radiological imaging will be performed 8 weeks ± 1 week, starting from date of randomization for the first 64 weeks, then every 16 weeks ± 1 week for the next 32 weeks, and then every 24 weeks ± 4 weeks thereafter.

SECONDARY OUTCOMES:
• To determine if AMG 386 plus PLD is superior to placebo plus PLD as measured by overall survival | weekly

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (93):
- United States (21):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Norwalk, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Evanston, Illinois
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, New York, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Abington, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Fort Sam Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Annandale, Virginia
  - Research Site, Green Bay, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, West Allis, Wisconsin
- Australia (8):
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Wahroonga, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Greenslopes, Queensland
  - Research Site, East Bentleigh, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Parkville, Victoria
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (8):
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Ieper
  - Research Site, Leuven
  - Research Site, Libramont
  - Research Site, Liège
  - Research Site, Namur
- Canada (2):
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
- Denmark (2):
  - Research Site, Copenhagen
  - Research Site, Herlev
- France (5):
  - Research Site, Amiens
  - Research Site, Avignon
  - Research Site, Lyon
  - Research Site, Poitiers
  - Research Site, Saint-Cloud
- Germany (12):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Hanover
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Tübingen
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Szeged
  - Research Site, Zalaegerszeg - Pozva
- Italy (5):
  - Research Site, Campobasso
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
- New Zealand (2):
  - Research Site, Grafton, Auckland
  - Research Site, Tauranga
- Poland (2):
  - Research Site, Bialystok
  - Research Site, Gdansk
- Research Site, Singapore, Singapore
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Prešov
- Switzerland (4):
  - Research Site, Aarau
  - Research Site, Chur
  - Research Site, Geneva
  - Research Site, Zurich
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (5):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Nottingham
  - Research Site, Poole

REFERENCES:
- [Background] Marth C, Vergote I, Scambia G, Oberaigner W, Clamp A, Berger R, Kurzeder C, Colombo N, Vuylsteke P, Lorusso D, Hall M, Renard V, Pignata S, Kristeleit R, Altintas S, Rustin G, Wenham RM, Mirza MR, Fong PC, Oza A, Monk BJ, Ma H, Vogl FD, Bach BA. ENGOT-ov-6/TRINOVA-2: Randomised, double-blind, phase 3 study of pegylated liposomal doxorubicin plus trebananib or placebo in women with recurrent partially platinum-sensitive or resistant ovarian cancer. Eur J Cancer. 2017 Jan;70:111-121. doi: 10.1016/j.ejca.2016.09.004. Epub 2016 Dec 1. PMID 27914241
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com